CLINICAL TRIAL: NCT00415935
Title: PRINTO (the Paediatric Rheumatology International Trials Organisation)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Child Health (Other)
Other Study IDs: 04RU01
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: methotrexate

SUMMARY:
A comparison of outcome in children with JIA who are in remission on MTX, when MTX is then stopped for either 6 or 12 months

ELIGIBILITY:
Inclusion Criteria:

* Any child with JIA who has gone into remission using methotrexate

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Wedderburn, Dr, Principal Investigator — Institute Of Child Health and Great Ormond Street Hospital
Locations (1):
- Rheumatology ICH, London, United Kingdom